CLINICAL TRIAL: NCT02899962
Title: LEO 90100 Twice Weekly Maintenance Regimen for Psoriasis Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0053-1004
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LEO 90100 aerosol foam (Active Comparator): Topical application twice weekly for 52 weeks
  Interventions: Drug: LEO 90100 aerosol foam
- LEO 90100 aerosol foam vehicle (Placebo Comparator): Topical application twice weekly for 52 weeks
  Interventions: Drug: LEO 90100 aerosol foam vehicle

INTERVENTIONS:
Drug: LEO 90100 aerosol foam — LEO 90100 aerosol foam twice weekly
  Arms: LEO 90100 aerosol foam
Drug: LEO 90100 aerosol foam vehicle — LEO 90100 aerosol foam vehicle twice weekly
  Arms: LEO 90100 aerosol foam vehicle

SUMMARY:
A phase 3 trial comparing the efficacy and safety of LEO 90100 aerosol foam with the aerosol foam vehicle used twice weekly as long-term maintenance therapy in subjects with psoriasis vulgaris.

A 12-month, international, multi-centre, randomised, vehicle controlled, double-blind, 2-arm, parallel group trial.

DETAILED DESCRIPTION:
After an initial 4-week period of once-daily treatment with open-label active LEO 90100 aerosol foam, subjects who qualify for randomisation will continue into a 52-week maintenance treatment period with twice-weekly application of randomised LEO 90100 aerosol foam / LEO 90100 aerosol foam vehicle.

If the subject experiences a relapse of psoriasis, the active lesions will be treated for 4 weeks with open-label active LEO 90100 aerosol foam.

ELIGIBILITY:
INCLUSION CRITERIA:

* A clinical diagnosis of psoriasis vulgaris for at least 6 months involving the trunk and/or limbs, amenable to treatment with maximum of 100 g of trial medication per week
* Psoriasis vulgaris on the trunk and/or limbs (excluding psoriasis on the genitals and skin folds) involving 2-30% of the body surface area (BSA)
* A target lesion/target location of at least 3 cm at its longest axis located on the body (i.e., not on the scalp, face or intertriginous areas), scoring at least 1 ('mild') for each of redness, thickness and scaliness, and at least 4 in total by the Investigator's Assessment of Severity of the Target Lesion/Location

For subjects participating in hypothalamic-pituitary-adrenal (HPA)-axis testing, furthermore:

* An extent of psoriasis vulgaris on trunk and/or limbs of disease severity (PGA) of at least 'moderate' affecting between 10 and 30% of the body surface area (BSA) excluding psoriatic lesions of genitals and skin folds at Visit 1.

EXCLUSION CRITERIA:

* Systemic treatment with biological therapies, whether marketed or not, with a possible effect on psoriasis vulgaris within the following time periods prior to Visit 1:

  * etanercept - within 4 weeks prior to Visit 1
  * adalimumab, infliximab - within 8 weeks prior to Visit 1
  * ustekinumab - within 16 weeks prior to Visit 1
  * secukinumab - within 12 weeks prior to Visit 1
  * other products - within 4 weeks/5 half-lives prior to Visit 1 (whichever is longer)
* Systemic treatment with all other therapies with a possible effect on psoriasis vulgaris (e.g. corticosteroids, retinoids, methotrexate, ciclosporin and other immunosuppressants) within 4 weeks prior to Visit 1
* Systemic treatment with apremilast within 4 weeks prior to Visit 1
* Psoralen combined with Ultraviolet A (PUVA) therapy within 4 weeks prior to Visit 1
* Ultraviolet B (UVB) therapy within 2 weeks prior to Visit 1
* Severe and/or extensive scalp psoriasis which, in the opinion of the investigator, requires treatment with potent or super-potent corticosteroids which will be prohibited during the trial

For subjects participating in HPA-axis testing, furthermore:

* Antidepressive medications within 4 weeks prior to Visit 1 or during the trial. Oestrogen therapy (including contraceptives), antidepressant medications and any other medication known to affect cortisol levels or HPA axis integrity within 4 weeks prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (58):
- United States (21):
  - Center for Dermatology Clinical Research, Fremont, California
  - Clinical Science Institute, Santa Monica, California
  - Colorado Medical Research Center, Denver, Colorado
  - International Dermatology Research, Miami, Florida
  - Arlington Dermatology, Arlington Heights, Illinois
  - Derm Research, Louisville, Kentucky
  - DermAssociates, Rockville, Maryland
  - Clarkston Skin Research, Clarkston, Michigan
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - Beyer Research, Kalamazoo, Michigan
  - Psoriasis Treatment Center of Central NJ, East Windsor, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Sadick Research Group, New York, New York
  - Skin Search of Rochester, Rochester, New York
  - UPMC Department of Dermatology, Pittsburgh, Pennsylvania
  - Rivergate Dermatology Clinical Research Center, Goodlettsville, Tennessee
  - The Skin Wellness Center, Knoxville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Clinical Trials of Texas, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Premier Clinical Research, Spokane, Washington
- Canada (12):
  - Dr. Chih-ho Hong Medical, Surrey, British Columbia
  - Pacific Dermaesthetics, Vancouver, British Columbia
  - Wiseman Dermatology Research, Winnipeg, Manitoba
  - Maritime Medical Research Centre, Bathurst, New Brunswick
  - Brunwick Dermatology Center, Fredericton, New Brunswick
  - CCA Medical Research, Ajax, Ontario
  - Dermatrials Research Incorporated, Hamilton, Ontario
  - The Guenther Dermatology Research Centre, London, Ontario
  - Lynderm Research, Markham, Ontario
  - SKiN Center for Dermatology, Peterborough, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Clinique du Dre Isabelle Delorme Inc, Québec, Quebec
- France (5):
  - C.H.U. de Saint-Etienne Service de Dermatologie, Saint-Etienne, Saint-Etienne
  - CHRU de Brest - Hôpital Morvan, Brest
  - C.H.U. de nice, Hôpital de l'Archet II, Service de Dermatologie-Vénérologie, Nice
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Centre Hospitalier de Valence, Valence
- Germany (9):
  - Klinik und Poliklinik für Dermatologie, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen (AöR), Klinik für Dermatologie, Essen
  - SRH Wald-Klinikum Gera, Gera
  - SCIderm GmbH, Hamburg
  - UKSH - Campus Lübeck, Lübeck
  - Michael Sebastian, Mahlow
  - LMU Poliklinik Derma & Allergo, München
  - Gemein. Weber & Crainic, Schweinfurt
- Poland (4):
  - Małopolskie Centrum Kliniczne, Krakow
  - NZOZ Med-laser, Lublin
  - Solumed, Poznan
  - Kliniczny Szpital Wojewódzki, Klinika Dermatologii, Rzeszów
- United Kingdom (7):
  - Wansford and Kings Cliffe Prac, Wansford, Cambridgeshire
  - Ashgate Medical Practice, Chesterfield, Derbyshire
  - Burbage Surgery, Burbage, Leicstershire
  - Albany House Medical Centre, Wellingborough, Northamptonshire
  - Sherbourne Medical Centre, Royal Leamington Spa, Warwickshire
  - Chapel Allerton Hospital, Leeds, West Yorkshire
  - Dermatopharmacology Department, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guenther L, Takhar A, Megna M, Sebastian M, Nyholm N, Thoning H, Levin LA. Impact of fixed-dose combination Cal/BD foam on the work productivity of patients with psoriasis: results from the 52-week randomized, double-blind, PSO-LONG trial. J Eur Acad Dermatol Venereol. 2022 Jul;36(7):1054-1063. doi: 10.1111/jdv.18053. Epub 2022 Mar 28. PMID 35297108
- [Derived] Lebwohl MG, Papp KA, Morch MH, Bernasconi MYJ, Warren RB. Long-Term Proactive Treatment of Plaque Psoriasis with Calcipotriene/Betamethasone Dipropionate Foam Prolongs Remission and Reduces Relapses Irrespective of Patient Baseline Characteristics. Dermatol Ther (Heidelb). 2021 Oct;11(5):1657-1665. doi: 10.1007/s13555-021-00585-x. Epub 2021 Aug 2. PMID 34339017
- [Derived] Stein Gold L, Alonso-Llamazares J, Lacour JP, Warren RB, Tyring SK, Kircik L, Yamauchi P, Lebwohl M; PSO-LONG Trial Investigators. PSO-LONG: Design of a Novel, 12-Month Clinical Trial of Topical, Proactive Maintenance with Twice-Weekly Cal/BD Foam in Psoriasis. Adv Ther. 2020 Nov;37(11):4730-4753. doi: 10.1007/s12325-020-01497-6. Epub 2020 Sep 23. PMID 32965655

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 722 subjects were screened of which 650 subjects were assigned to treatment with LEO 90100 open-label phase. Subjects did not progress from screening due to adverse event=1, lost to follow-up=2, other reasons=2, screening failures=52, and withdrawal by subject=15. All 650 subjects were exposed to LEO 90100 during the open-label phase
Groups:
- Open-label LEO 90100: In the open-label phase, LEO 90100, an aerosol foam formulation containing calcipotriol 50 mcg/g (as hydrate) and betamethasone 0.5 mg/g (as dipropionate) was applied once daily on the body for 4 weeks.
- Maintenance LEO 90100: In the maintenance phase, subjects from open-label phase who achieved treatment success according to Physician's Global Assessment of disease severity (clear or almost clear with 2-step improvement) were randomised to receive LEO 90100 twice weekly for 52 weeks. In case of relapse (psoriasis which was mild, moderate or severe according to PGA), rescue medication was applied. Rescue medication was LEO 90100 applied once daily on the body for 4 weeks.
- Maintenance Vehicle: In the maintenance phase, subjects from open-label phase who achieved treatment success according to Physician's Global Assessment of disease severity (clear or almost clear with 2-step improvement) were randomised to receive vehicle twice weekly for 52 weeks. In case of relapse (psoriasis which was mild, moderate or severe according to PGA), rescue medication was applied. Rescue medication was LEO 90100 applied once daily on the body for 4 weeks.
Period: Open-label Phase
Arm/Group | Open-label LEO 90100 | Maintenance LEO 90100 | Maintenance Vehicle
Started | 650 | 0 | 0
Completed | 623 | 0 | 0
Not Completed | 27 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Lost to Follow-up | 9 | 0 | 0
Not completed — Other reasons | 9 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0
Period: Maintenance Phase
Arm/Group | Open-label LEO 90100 | Maintenance LEO 90100 | Maintenance Vehicle
Started | 0 | 272 | 273
Completed | 0 | 131 | 120
Not Completed | 0 | 141 | 153
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 20 | 16
Not completed — Lost to Follow-up | 0 | 12 | 14
Not completed — Other reasons | 0 | 9 | 13
Not completed — Not achieve treatment success after Wk 4 | 0 | 3 | 2
Not completed — Not clear/almost clear after rescue med | 0 | 65 | 70
Not completed — Withdrawal by Subject | 0 | 30 | 36

BASELINE CHARACTERISTICS:
Population: Included all subjects exposed to LEO 90100 at the start of open-label phase
Groups:
- LEO 90100 Open-label Phase: LEO 90100, an aerosol foam formulation containing calcipotriol 50 mcg/g (as hydrate) and betamethasone 0.5 mg/g (as dipropionate) was applied once daily on the body for 4 weeks.
Arm/Group | LEO 90100 Open-label Phase
Number analyzed (Participants) | 650
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.8 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226
  Male | 424
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 75
  Not Hispanic or Latino | 568
  Unknown or Not Reported | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data available only from 635 subjects
  Participants
    Race: number analyzed (Participants) | 635
    Race: White | 584
    Race: Asian | 37
    Race: Black or African American | 9
    Race: Native Hawaiian or Other Pacific Islander | 4
    Race: American Indian or Alaska Native | 1
Region of Enrollment [Number; unit: participants]
  Canada | 163
  United States | 228
  Poland | 60
  United Kingdom | 79
  France | 61
  Germany | 59
PGA [Count of Participants; unit: Participants] — The investigator was to grade the severity of psoriasis of the trunk and limbs using the 5-point scale Physician's global assessment of the disease severity:
  Clear = 0; Almost clear = 1; Mild = 2; Moderate = 3; Severe = 4
  Participants
    Mild | 83
    Moderate | 509
    Severe | 58

OUTCOME MEASURES:

1. Primary Outcome: Time to First Relapse
Description: Time to first relapse (at least 'mild' according to the Physician's Global Assessment of disease severity [PGA]). The investigator was to grade the severity of psoriasis of the trunk and limbs using Physician's global assessment of disease severity 5-point scale: Clear = 0; Almost clear = 1; Mild = 2; Moderate = 3; Severe = 4
Time Frame: From Randomisation (Week 4) until first relapse or End of Treatment (Week 56 or early withdrawal)
Population: Full analysis set: included all subjects randomised who had treatment success at randomisation, defined as PGA score of 'clear' or 'almost clear' with at least a 2-grade improvement from baseline
Measure: Median (95% Confidence Interval); unit: days
Groups:
- LEO 90100 Aerosol Foam: Topical application of LEO 90100 aerosol foam twice weekly for 52 weeks
- LEO 90100 Aerosol Foam Vehicle: Topical application of LEO 90100 aerosol foam vehicle twice weekly for 52 weeks
Arm/Group | LEO 90100 Aerosol Foam | LEO 90100 Aerosol Foam Vehicle
Number analyzed (Participants) | 256 | 265
days | 56 [34 to 59] | 30 [29 to 31]
Statistical Analysis 1: Comparison: LEO 90100 Aerosol Foam vs LEO 90100 Aerosol Foam Vehicle; All randomized subjects were considered for statistical analysis; Test type: Superiority — The primary endpoint was time to first relapse during the maintenance phase. This was calculated as the number of days from randomisation to the day where the subject had the first relapse confirmed. For subjects who either did not encounter a relapse or were withdrawn from the trial, the number of days was treated as a censored observation at the day of end of trial visit; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.47 to 0.69] — Estimates are obtained from a proportional hazards model with treatment group,pooled trial site,disease severity at maintenance baseline (Week 4; determined by PGA) as factors

2. Secondary Outcome: Proportion of Days in Remission During the Maintenance Phase
Description: Remission defined as 'clear' or 'almost clear' according to the PGA. The investigator was to grade using a global assessment of the disease severity of psoriasis of the trunk and limbs using the PGA 5-point scale: Clear = 0; Almost clear = 1; Mild = 2; Moderate = 3; Severe = 4
Time Frame: From Randomisation (Week 4) until End of Treatment (Week 56 or early withdrawal)
Measure: Mean (Standard Deviation); unit: Proportion of days
Arm/Group | LEO 90100 Aerosol Foam | LEO 90100 Aerosol Foam Vehicle
Number analyzed (Participants) | 256 | 265
Proportion of days | 70.2 (21.7) | 60.8 (20.1)
Statistical Analysis 1: Comparison: LEO 90100 Aerosol Foam vs LEO 90100 Aerosol Foam Vehicle; The number of days in remission was calculated as the sum of days where the subject was in remission periods. The proportion of days in remission was calculated as the number of days in remission divided by the length of the maintenance phase in days; Test type: Superiority; p < 0.001, ANOVA; Factors adjusted for in the ANOVA model were treatment group, pooled trial site, and disease severity at maintenance baseline (PGA); Mean Difference (Net) = 0.11, 95% CI 2-sided [0.08 to 0.14] — Multiple imputation of data for withdrawn subjects was done using 100 imputations and depended on whether the subject's reason for withdrawal potentially was related to treatment. Length of the maintenance phase was assumed to be 52 weeks (364 days)

3. Secondary Outcome: Number of Relapses During the Maintenance Phase
Description: Defined as number of 4-week periods with use of once-daily rescue investigational medicinal product
Time Frame: From Randomisation (Week 4) until End of Treatment (Week 56)
Measure: Mean (Standard Deviation); unit: relapses
Arm/Group | LEO 90100 Aerosol Foam | LEO 90100 Aerosol Foam Vehicle
Number analyzed (Participants) | 256 | 265
relapses | 2.0 (1.7) | 3.1 (2.2)
Statistical Analysis 1: Comparison: LEO 90100 Aerosol Foam vs LEO 90100 Aerosol Foam Vehicle; Test type: Superiority; p < 0.001, Poisson regression; Rate ratio = 0.54, 95% CI 2-sided [0.46 to 0.63] — The number of relapses was analysed using a Poisson regression model with treatment group,pooled sites,disease severity at maintenance baseline as factors, subject as random effect, and time at risk as an offset

ADVERSE EVENTS:
Time Frame: 4 weeks during the open-label phase and 52 weeks during the maintenance phase and 8 weeks during the safety follow-up
Description: All adverse events were reported by the subjects or observed by the investigators were recorded
Groups:
- LEO 90100 Aerosol Foam Open-label: Topical application once daily for 4 weeks
  LEO 90100 aerosol foam open-label
Arm/Group | LEO 90100 Aerosol Foam Open-label | LEO 90100 Aerosol Foam | LEO 90100 Aerosol Foam Vehicle
All-Cause Mortality (participants affected / at risk) | 0/650 | 0/272 | 1/273
Serious Adverse Events (participants affected / at risk) | 4/650 | 14/272 | 11/273
Other Adverse Events (participants affected / at risk) | 47/650 | 83/272 | 87/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 90100 Aerosol Foam Open-label (N=650) | LEO 90100 Aerosol Foam (N=272) | LEO 90100 Aerosol Foam Vehicle (N=273)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (4)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arterial stenosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 90100 Aerosol Foam Open-label (N=650) | LEO 90100 Aerosol Foam (N=272) | LEO 90100 Aerosol Foam Vehicle (N=273)
Vitamin D deficiency (Metabolism and nutrition disorders) | 36 (36) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 16 (17) | 15 (24)
Nasopharyngitis (Infections and infestations) | 7 (7) | 22 (23) | 19 (24)
Influenza (Infections and infestations) | 2 (2) | 7 (7) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 6 (6)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 5 (5)
Sinusitis (Infections and infestations) | 2 (2) | 5 (5) | 2 (3)
Gastroenteritis (Infections and infestations) | 3 (3) | 4 (4) | 2 (2)
Folliculitis (Infections and infestations) | 2 (2) | 4 (4) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
Rebound psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 12 (12)
Psoriasis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 7 (7)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (7) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 5 (5) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 4 (4)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3)
Sciatica (Nervous system disorders) | 0 (0) | 4 (4) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 6 (6) | 4 (4) | 3 (3)
Cataract (Eye disorders) | 0 (0) | 3 (4) | 0 (0)
Chest pain (General disorders) | 1 (1) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma acknowledges the investigators' right to publish the entire results of the study, irrespective of outcome. LEO Pharma retains the right to have any publication submitted to LEO Pharma for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO Pharma.

DOCUMENTS (2):
  • Study Protocol (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT02899962/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT02899962/SAP_001.pdf